CLINICAL TRIAL: NCT00602043
Title: A Phase 2 Study of [18F] Fluoroestradiol (FES) as a Marker of Hormone Sensitivity of Metastatic Breast Cancer
Brief Title: F-18 16 Alpha-Fluoroestradiol-Labeled Positron Emission Tomography in Predicting Response to First-Line Hormone Therapy in Patients With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2009-00270; NCI-2009-00270 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB #6590; CDR0000584077; UWCC-6590; IRB #6590 (Other: University of Washington Medical Center); 8052 (Other: CTEP)
Record Dates: First submitted 2008-01-23; First posted 2008-01-28 (Estimated); Results first posted 2014-12-25 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Estrogen Receptor-positive Breast Cancer; Progesterone Receptor-negative Breast Cancer; Progesterone Receptor-positive Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

ARMS (1):
- Diagnostic (FES) (Experimental): Patients undergo [^18F] FES PET scan. Patients also undergo standard clinical fludeoxyglucose F 18 (FDG)-PET or FDG-PET/CT scan up to 14 days prior to [^18F] FES PET scan.
  Interventions: Radiation: F-18 16 alpha-fluoroestradiol; Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography; Procedure: computed tomography; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: F-18 16 alpha-fluoroestradiol — Undergo [^18F] FES PET
  Other Names: F-18 FES; fluorine-18 16 alpha-fluoroestradiol
Radiation: fludeoxyglucose F 18 — Undergo standard clinical FDG PET/CT
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Undergo [^18F] FES PET
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: positron emission tomography — Undergo standard clinical FDG PET/CT
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo standard clinical FDG PET/CT
  Other Names: tomography, computed
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well F-18 16 alpha-fluoroestradiol (FES) imaging works in predicting response to first-line hormone therapy in women with hormone receptor-positive metastatic breast cancer. Diagnostic procedures, such as FES imaging, may help predict how well patients will respond to hormone therapy and may help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the ability of [^18F] FES positron emission tomography (PET) or PET/computed tomography (CT) uptake at the level of standard uptake value (SUV) < 1.5 to predict overall response (OR) to first line endocrine therapy for metastatic breast cancer.

SECONDARY OBJECTIVES:

I. Evaluate the independent role of [^18F] FES in predicting response and time to progression in patients treated with first-line endocrine therapy for metastatic breast cancer.

II. Examine the role of [^18F] FES in predicting OR or clinical benefit (CB), in concert with tissue assay of levels of estrogen receptor (ER) messenger ribonucleic acid (mRNA) measured using quantitative polymerase chain reaction (PCR), and semi-quantitative interpretation of estrogen receptor (ER), progesterone receptor (PgR), androgen receptor (AR), and human epidermal growth factor-2 (HER2), in addition to serial measures of hormone levels in plasma.

III. Evaluate the relationships among [^18F] FES, semi-quantitative ER from immunohistochemistry (IHC), and ER mRNA as measured by quantitative PCR.

IV. Document the safety profile of [^18F] FES PET in newly diagnosed patients with metastatic breast cancer.

V. Evaluate FES SUV < 1.5 as the optimal cutpoint for predicting OR to first-line endocrine therapy for metastatic breast cancer.

VI. Estimate the rate of [^18F] FES SUV < 1.5 in newly diagnosed metastatic breast cancer patients planning a course of endocrine therapy.

OUTLINE:

Patients undergo [^18F] FES PET scan. Patients also undergo standard clinical fludeoxyglucose F 18 (FDG)-PET or FDG-PET/CT scan up to 14 days prior to [^18F] FES PET scan.

After completion of study treatment, patients are followed up for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have pathologically confirmed invasive breast cancer with clinical, radiographic and/or pathologic evidence of stage IV disease; patients must have tissue blocks available from biopsy of at least one site of metastatic disease and/or from diagnosis of their primary breast cancer
* Disease may be measurable (by Response Evaluation Criteria in Solid Tumors [RECIST] criteria) or non-measurable but must be present in at least one non-liver site and imageable on FDG PET scan; in patients with non-measurable disease by RECIST criteria, one of the following may be used to assess and follow disease: MUC-1 antigen level (either cancer antigen [CA] 27.29 or carcinoembryonic antigen [CEA]) > 2 x upper limit of normal (ULN), Circulating tumor cell assay > 5, or FDG-PET SUV > 2.5 in purely lytic lesions; elevated tumor markers alone are insufficient
* No prior endocrine therapy for breast cancer or

  * Off adjuvant endocrine therapy for > 6 months or
  * Greater than 2 years of a single adjuvant endocrine therapy at the time of first recurrence and plan to change to alternate endocrine therapy; use of tamoxifen must be discontinued 6-8 weeks prior to entrance into the study
* Prior chemotherapy regimens in the adjuvant or neoadjuvant setting are allowed
* Women treated with adjuvant LHRH (luteinizing hormone-releasing hormone) analog are eligible
* Be assessed for menopausal status; for study purposes, postmenopausal is defined as:

  * A prior documented bilateral oophorectomy, or
  * A history of at least 12 months without spontaneous menstrual bleeding, or
  * Age 60 or older with a prior hysterectomy without oophorectomy, or
  * Age less than 60 with a prior hysterectomy without oophorectomy (or in whom the status of the ovaries is unknown), with a documented follicle stimulating hormone (FSH) level demonstrating confirmatory elevation in the postmenopausal range for the lab
* Premenopausal patients must have a baseline FSH, and estradiol levels to determine menopausal status; measures will be repeated at 3-6 months to confirm menopausal status
* Patients must be positive for estrogen receptor (ER) and may or may not be positive for progesterone receptor (PgR) by IHC in the primary tumor and/or metastatic site; the pathology report for assay of ER will be reviewed by one of the investigators prior to enrollment, the study pathologist will review the pathology report if necessary for determination of study eligibility
* Tumor HER2/neu expression must be determined prior to study enrollment; assessment may be by fluorescence in situ hybridization (FISH) assay or by immunohistochemistry (ICC); if determination is intermediate by ICC, FISH must be performed
* Life expectancy > 16 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1,000
* Platelet count >= 50,000
* Hemoglobin within normal limits (WNL) for the institution
* Serum creatinine =< 1.5 x institutional ULN (IULN) and estimated creatinine clearance > 50 mL/min using the Cockroft-Gault formula
* Bilirubin =< 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT)/ serum glutamic pyruvate transaminase (SGPT) =< 1.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Patients must be planning a course of endocrine therapy with one of the following: tamoxifen +/- ovarian suppression, aromatase inhibitor +/- fulvestrant (with ovarian suppression in pre-menopausal patients) or fulvestrant alone
* After entry into the study, patients are expected to be followed for at least 6 months after the injection of [^18F] FES
* Have a negative pregnancy test within 7 days prior to registration if of childbearing potential
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer from which the patient has been disease-free for 5 years
* Be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific screening procedures
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Patients with a history of prior endocrine therapy for metastatic disease are NOT eligible; adjuvant endocrine therapy for < 2 years total or discontinued less than 6 months before first disease recurrence also excludes the patient
* Patients with disease in the liver only are NOT eligible for the study
* Patients who are HER2/neu positive disease and planning to undergo HER2-directed therapy (trastuzumab or lapatinib) are NOT eligible for the study
* Pregnant or lactating; women of childbearing potential with either a positive or no pregnancy test at baseline are excluded
* Visceral crisis characterized by rapidly progressive hepatic or lymphangitic lung metastases
* History of uncontrolled seizures, central nervous system disorders, or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent
* Any other life-threatening illness (e.g., serious, uncontrolled concurrent infection or clinically significant cardiac disease - congestive heart failure, symptomatic coronary artery disease, cardiac arrhythmia not well controlled with medication)
* Unwillingness to give informed consent
* Medically unstable as judged by the patient's physician
* Psychological, familial, sociological, or geographical conditions which do not permit compliance with the study protocol
* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals; patients with significant drug or other allergies or autoimmune diseases may be enrolled at the investigator's discretion
* Patient weight greater than 400 lbs (exceeds weight limit for tomograph table)
* Uncontrolled diabetes mellitus (fasting glucose > 200 mg/dL)
* Adult patients who require monitored anesthesia for PET scanning

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet F Eary, MD, Principal Investigator — Department of Radiology, University of Alabama, Birmingham, AL; David A Mankoff, MD, PhD, Study Director — University of Pennsylvania
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Result] Peterson LM, Kurland BF, Schubert EK, Link JM, Gadi VK, Specht JM, Eary JF, Porter P, Shankar LK, Mankoff DA, Linden HM. A phase 2 study of 16alpha-[18F]-fluoro-17beta-estradiol positron emission tomography (FES-PET) as a marker of hormone sensitivity in metastatic breast cancer (MBC). Mol Imaging Biol. 2014 Jun;16(3):431-40. doi: 10.1007/s11307-013-0699-7. Epub 2013 Oct 30. PMID 24170452

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (FES): Patients undergo [^18F] FES PET scan. Patients also undergo standard clinical fludeoxyglucose F 18 (FDG)-PET or FDG-PET/CT scan up to 14 days prior to [^18F] FES PET scan.
  Patients begin clinically indicated endocrine therapy.
  Patients are followed-up to determine response on the therapy for 6 months using clinical exams, tumor marker assays, conventional imaging and standard clinical FDG PET/CT.
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Diagnostic (FES)
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | First Line Endocrine Therapy for a Stage IV Disease
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Patients were expected to start endocrine therapy within 2 weeks of the FES PET scan. Response assessment was evaluated at 3 and 6 months. For patients with at least one site of measurable disease [per response evaluation criteria in solid tumors (RECIST, version 1.1)], size-based response criteria were used to assess response.
  For patients without disease evaluable by RECIST 1.1, largely patients with bone-dominant metastatic breast cancer, serial FDG PET scanning was used to determine response. A decline in the FDG PET SUV (standard uptake value) of 30% or more was considered as response and an increase of 20% or more was considered to be progressive disease (PD).
  The initial (baseline) FES uptake was compared to clinical benefit (PD versus other outcome at 6 months).
Time Frame: Up to 6 months
Measure: Number; unit: patients with progressive disease
Groups:
- Diagnostic FES: Average FES SUVmean >1.5, no Negative Sites: Patients undergo [^18F] FES PET scan. Patients also undergo standard clinical fludeoxyglucose F 18 (FDG)-PET or FDG-PET/CT scan up to 14 days prior to [^18F] FES PET scan.
  Patients begin clinically indicated endocrine therapy.
  Patients are followed-up to determine response on the therapy for 6 months using clinical exams, tumor marker assays, conventional imaging and standard clinical FDG PET/CT.
  This group represents patients who had positive FES uptake at all disease sites on the baseline diagnostic FES PET scan.
  laboratory biomarker analysis: Correlative studies
- Diagnostic FES: Patients With FES Negative Sites of Disease: Patients undergo [^18F] FES PET scan. Patients also undergo standard clinical fludeoxyglucose F 18 (FDG)-PET or FDG-PET/CT scan up to 14 days prior to [^18F] FES PET scan.
  Patients begin clinically indicated endocrine therapy.
  Patients are followed-up to determine response on the therapy for 6 months using clinical exams, tumor marker assays, conventional imaging and standard clinical FDG PET/CT.
  This group represents patients who had some or all disease sites negative for FES uptake on the baseline diagnostic FES PET scan.
Arm/Group | Diagnostic FES: Average FES SUVmean >1.5, no Negative Sites | Diagnostic FES: Patients With FES Negative Sites of Disease
Number analyzed (Participants) | 13 | 3
patients with progressive disease | 5 | 2

2. Secondary Outcome: Number of Participants With Clinical Benefit
Description: FES SUV prior to endocrine treatment (dichotomized and as a continuous predictor) will also be tested as predictor of clinical benefit.
  Patients were expected to start endocrine therapy within 2 weeks of the FES PET scan. Response assessment was evaluated at 3 and 6 months.
  The initial (baseline) FES uptake was compared to clinical benefit (PD versus other outcome at 6 months).
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic FES: Average FES SUVmean >1.5, no Negative Sites | Diagnostic FES: Patients With FES Negative Sites of Disease
Number analyzed (Participants) | 13 | 3
Participants | 8 | 0

3. Secondary Outcome: Time to Progression
Description: FES SUV prior to endocrine treatment (dichotomized and as a continuous predictor) will also be tested as predictor of time to progression. Analysis will be conducted using (respectively) logistic regression and Cox proportional hazards regression. This will include univariate analysis of FES and other predictive measures (ER/PgR expression, serum sex steroid levels), followed by an exploratory multivariate analysis combining FES SUV with other measures showing predictive capability univariate analysis.
Time Frame: Up to 6 months
Measure: Median (Full Range); unit: months
Groups:
- Diagnostic (FES): Average FES SUVmean >1.5, no Negative Sites: Patients undergo [^18F] FES PET scan. Patients also undergo standard clinical fludeoxyglucose F 18 (FDG)-PET or FDG-PET/CT scan up to 14 days prior to [^18F] FES PET scan.
  Patients begin clinically indicated endocrine therapy.
  Patients are followed-up to determine response on the therapy for 6 months using clinical exams, tumor marker assays, conventional imaging and standard clinical FDG PET/CT.
  This group represents patients who had positive FES uptake at all disease sites on the baseline diagnostic FES PET scan.
Arm/Group | Diagnostic (FES): Average FES SUVmean >1.5, no Negative Sites | Diagnostic FES: Patients With FES Negative Sites of Disease
Number analyzed (Participants) | 5 | 2
months | 4.9 [2.1 to 6.0] | 2.2 [1.2 to 3.3]

4. Secondary Outcome: Correlation of FES Uptake With ER Assays
Description: Graphical and numerical studies of bivariate relationships will be examined, as well as factors (i.e., tumor size, tumor location, patient age) to explain concurrence, lack of concurrence, and sources of measurement error for measurements of ER function.
Time Frame: Up to 6 months
Population: Data were not collected due to variations in reporting methods for ER assays.
Arm/Group | Diagnostic (FES)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Diagnostic (FES)
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less